CLINICAL TRIAL: NCT04367441
Title: A Study of Single Dose Escalation, Randomized, Double Blinded, Placebo Controlled to Investigate the Tolerability, Safety Profiles, Pharmacokinetic of Recombinant Humanized Anti-IL17A Monoclonal Antibody Injection in Healthy Subjects
Brief Title: Randomized, Double Blinded, Placebo Controlled, Single Dose Escalation Study of 608 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ -608- Psoriasis-I-01
Record Dates: First submitted 2020-04-25; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 608 (Experimental): 8mg, 20mg, 40mg, 80mg, 120mg, 160mg, 200mg
  Interventions: Drug: 608
- Placebo (Placebo Comparator): 20mg, 40mg, 80mg, 120mg, 160mg, 200mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 608 — recombinant humanized anti-IL17A monoclonal antibody injection
  Arms: 608
Drug: Placebo — auxiliary material of 608 include histidine, histidine hydrochloride, sucrose and polysorbate 80
  Arms: Placebo

SUMMARY:
This is a first-in-human, phase 1, single-center, randomized, double blinded, placebo-controlled, single dose-escalation study to evaluate the safety, tolerability, PK, of 608 following subcutaneous injection in healthy subjects.

DETAILED DESCRIPTION:
The study will consist of a 14-days screening period (-14~-1 days); an observation period (7-14 days) and the follow-up period (71-91days); Subjects will be randomly assigned to seven group.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 45 years;
* Good health status (no significant clinical symptoms and signs and no clinical significance of abnormal laboratory test).
* The body weight no less than 50 kg for male subjects and no less than 45 kg for female subjects. Body mass index (BMI) = weight (kg)/square of height, ranging from 19-26kg/m2 (including the critical value)
* Voluntary written informed consent;
* Being able to complete the study according to the requirements in the study protocol
* The person who have undergone surgical treatment have fully recovered

Exclusion Criteria:

* Allergic constitution or history of allergy to two or more substances; Known hypersensitivity to any biotherapy; Allergy to rubber or latex; Allergy to study drug or any components of study drug by investigator assessment
* Participation in any other clinical study about drugs or medical instruments within 3 months prior to enroll, or subjects currently included in the study which are not scientifically or medically compatible with this study
* Use of any medicine within 5 half-lives or less than 4 weeks prior to enroll (the longer of the two shall prevail)
* Participation in any IL-17 antagonists at any time
* Used vaccination or participation in any other clinical vaccination study within 12 weeks prior to enroll, or plan to use vaccine during the study or within 12 months after the study
* Any major surgery within 8 weeks prior to enroll, or requiring such surgery during the study
* Having history of any clinically significant diseases, including but not limited to digestive system, cardiovascular system, respiratory system, urinary system, musculoskeletal system, endocrine system, nerves and mental system, hematological system, Immune diseases, abnormal metabolism, etc
* History of or current Inflammatory Bowel Disease
* Loss or donation of blood ≥200mL within 12 weeks prior to enroll, or receiving blood transfusion in recent 8 weeks; or plan to donate blood during the study
* Positive HIV antibody or positive treponema pallidum serum specific antibody;
* Positive hepatitis B surface antigen, or positive hepatitis B core antibody and negative hepatitis B surface antibody
* Positive hepatitis C antibody
* History of or current lymphatic proliferative disease; Sign or symptom of lymphatic proliferative disease; History of or current malignant tumor
* Serious infection (e.g., pneumonia, cellulitis) or varicella-zoster virus infection, hospitalization, infection using antibiotics by intravenous injection within 12 weeks prior to enroll; serious bone and joint infection witn 24 weeks prior to enroll; or happened artificial joint infections; any infection within 7 days (include chronic or local infection ,such as a local skin infection); or history of recurrent infections and prone to infections of the basic diseases ((including but not limited to herpes zoster virus (> 1 time) and herpes simplex virus infection); history of any immunological injuries(pneumocystis pneumonia, histoplasmosis, or coccidioidomycosis);
* Having clinical evidence of active tuberculosis or suspected for active TB, or previous evidence of active TB but not received appropriate treatment or missing records; or latent tuberculosis infection at screening;
* Known immune deficiency; or the subject with weakened immune system may have unacceptable risk if participating in this study
* Pregnant, nursing, or planning pregnancy within 6 months(women) or planning to donate sperm or egg; pregnancy test positive; not use effective contraception (details for appendix 5) or the partner of the men subject planned to have a baby within 6 months;
* History of definite neurological or psychiatric disorders:such as epilepsy;
* History of alcohol or substance abuse with 14 units of alcohol per week within 6 months (1 unit =12 ounce or 360mL beer/1.5 ounce or 45ml liquor with 40% alcohol/5 ounce or 150mL wine); positive of alcohol or substance abuse test;
* Smoking more than 5 per day within 6 months prior to enroll
* Chronic overdose of tea, coffee, or caffeinated beverages within 3 months (average more than 8 cups per day, 1 cup=250mL);having any food or beverages with alcohol / caffeine within 48 hours prior to administration (such as coffee, strong tea, cocoa, chocolate and so on); having any food or beverages with rich grapefruit, grapefruit juice or others effect on absorption distribution, metabolism, excretion;
* insufficient understanding of the content and unwilling to comply with arrangement and other sides do not meet the inclusion criteria
* Any other conditions, the subject was inappropriate to participate in the study by investigators evaluated (for example, weak or having a disease that prevents the subjects from completing the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
AE/SAEs | From baseline through overall study (follow-up period: the arm of 8mg, 20mg,40mg with 71 days; 80mg, 120mg,160mg, 200mg with 91 days)
  Incidence of treatment emergent AE/SAEs

SECONDARY OUTCOMES:
Cmax | From baseline through 71days/91day
  Maximum observed concentration (Cmax) of 608
Tmax | From baseline through 71days/91day
  Time to Reach the Maximum Concentration After Drug Administration (Tmax) in 608 group
AUClast | From baseline through 71days/91day
  Area Under the Serum Concentration-time Cure From Time Zero to the Time of Last Quantifiable Concentration (AUClast) in 608 group.
AUCinf | From baseline through 71days/91day
  Area Under the Serum Concentration-time Curve From Time Zero to (AUCinf) in 608 group.
CL | From baseline through 71days/91day
  Systemic Clearance From Serum Following Intravenous Administration (CL) in 608 group
Vd | From baseline through 71days/91day
  Apparent volume of distribution (Vd) in 608 group
T1/2 | From baseline through 71days/91day
  Terminal Elimination Half-life (T1/2) in 608 group
MRT | From baseline through 71days/91day
  Mean residence time (MRT) in 608 group
λz | From baseline through 71days/91day
  Apparent terminal elimination rate constant (λz)in 608 group.
Percentage of Participants With Anti-608 Antibodies | From baseline through 71days/91day.
  Percentage of participants with treatment-emergent positive anti-608 antibodies and Neutralizing antibody;

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Clinical Center (Shanghai), Zhujing, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided